CLINICAL TRIAL: NCT05866133
Title: Relationship of Addictions to Obesity, Physical Activity and Vascular Ageing in Young Adults
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fundacion para la Investigacion y Formacion en Ciencias de la Salud (Other)
Collaborators: Castilla-León Health Service (Other); Instituto de Investigación Biomédica de Salamanca (Other)
Responsible Party: Sponsor
Other Study IDs: GRS 2500/B/22; IBYE22/00003 (Other Grant/Funding Number: IBSAL)
Record Dates: First submitted 2023-04-28; First posted 2023-05-19 (Actual); Last update posted 2023-05-19 (Actual); Status verified 2023-04

CONDITIONS: Drug Addiction; Technology Addiction; Young Adult
Keywords: Lifestyles; Vascular ageing; Obesity
MeSH Terms: conditions — Substance-Related Disorders; Technology Addiction; Obesity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Young people with addiction: Both behavioural and drug addiction will be assessed. Participants with scores consistent with an addiction will be included in this group.
- Young people without addiction: Both behavioural and drug addiction will be assessed. Participants with scores not consistent with an addiction will be included in this group.

SUMMARY:
This is a cross-sectional observational study whose objective is to analyse the relationship between behavioural addictions and drug addictions with obesity, physical activity, sedentary lifestyle, arterial stiffness and vascular ageing in young adults, since many of the lifestyles of adulthood are established early in life, and it is easier to prevent them before they start than to achieve their abandonment once they are established as unhealthy lifestyles

DETAILED DESCRIPTION:
Behavioural addictions. Brief Questionnaire of Pathological Gambling (CBJP), Lie/Bet scale, Compulsive Internet Use Scale (CIUS), Smartphone Dependence and Addiction Scale (EDAS-18), Questionnaire of Experiences Related to Video Games (CERV). Drug addictions: Alcohol, Smoking and Substance Involvement Screening Test (ASSIST V3.0), Drug Abuse Screening Test (DAST-20), Alcohol Use Disorders Identification Test (AUDIT) and Fagerström test. Obesity and body composition: Weight, height, waist circumference, hip circumference and Inbody 230®. Diet: Mediterranean Diet Adherence Questionnaire. Physical activity: International Physical Activity Questionnaire (IPAQ), Actigraph GTX3 accelerometer and Marshall questionnaire. Analysis of vascular structure and function and target organ lesions. Pulse wave analysis (PWA) and femoral carotid pulse wave velocity (VOPcf) (Sphygmocor System). Cardio Ankle Vascular Index (CAVI), ankle-ankle pulse wave (VOPbt) and ankle-ankle index (ABI) (Vasera VS-2000®). Retinal vascular injury (TOPCON TRC NW 200). Cardiac lesion (General electric 5000). Kidney Injury: analytical variables. Brain Injury: Montreal Cognitive Assessment (MoCA). Vascular ageing (VOPcf and VOPbt). Other variables. Basal glycaemia, HbA1c. TSH, lipid profile, creatinine and creatinine albumin index and Vit D. Measurement of blood pressure and drug consumption.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 18 and 34 years of age who agree to participate in the study and do not meet any exclusion criteria.

Exclusion Criteria:

* Subjects who are terminally ill, who are unable to travel to health centres for the corresponding examinations, and who do not sign informed consent.

Ages: 18 Years to 34 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Urban population assigned to the health area of Salamanca. By means of stratified random sampling by age and sex groups with replacement, based on the individual health card (TIS), subjects aged between 18 and 34 years will be selected.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-04-17 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-03-30 (Estimated)

PRIMARY OUTCOMES:
Pulse wave velocity | 1 year
  Measurement by SphygmoCor (meters/seg)

SECONDARY OUTCOMES:
Cardio Ankle Vascular Index (CAVI) | 1 year
  It will be determined using the Vasera VS-2000® device (not units)
Pathological gambling | 1 year
  Brief Questionnaire on Pathological Gambling (CBJP), with 4 dichotomous items (yes/no) referring to gambling habits, feelings of guilt, inability to give up gambling and use of household money for gambling. It is considered pathological from 2 points onwards. Also, Lie/Bet scale will also be used. It consists of two items, one of them referring to lying and the other to gambling, and will be considered problematic if both items are answered positively.
Internet use | 1 year
  Compulsive Internet Use Scale (CIUS). It consists of 14 questions with a 5-point Likert scale for the answer. The cut-off point is 28.
Compulsive use of mobile phones | 1 year
  Smartphone Dependence and Addiction Scale (EDAS-18). It consists of 18 questions with a 5-point Likert scale for the answer. Average scores: No dependence: ≤ 2.23; dependence: between 2.24 and 3.5; addiction: ≥ 3,6
Videogames use | 1 year
  Video Game Related Experiences Questionnaire (VREQ), with two dimensions: negative consequences and avoidance. It consists of 17 questions with a 4-point Likert scale for the answer. The cut-off point is 26 points.
Use or abuse of alcohol, tobacco and illegal drugs | 1 year
  Alcohol, Smoking and Substance Involvement Screening Test (ASSIST V3.0), with 8 items in relation to the consumption of 9 substances, categorised into three risk levels: low (0-3 points), moderate (4-26 points) and high (more than 27 points).
Problem drug use | 1 year
  Drug Abuse Screening Test (DAST-20), 20 questions with dichotomous answers (Yes/No) and a cut-off point of 5
Excessive alcohol consumption | 1 year
  Alcohol Use Disorders Identification Test (AUDIT), with 10 questions, allows to identify: risky use (8-15 points), harmful use (16-19 points) and dependence (more than 20 points)
Nicotine dependence | 1 year
  Fagerström test. With six questions it classifies into mild (less than 4 points), moderate (4-6 points) or severe dependence (more than 7 points).
Waist and hip circumference | 1 year
  The waist and hip circumference shall be measured with a tape measure (cm).
Body composition | 1 year
  The analysis of body composition shall be carried out with the impedance-meter Inbody 230® (kg).
International Physical Activity Questionnaire (IPAQ) | 1 year
  Physical activity measurement using the International Physical Activity Questionnaire (IPAQ) (min/day)
Accelerometer | 1 year
  Physical activity measurement using actigraph GTX3 accelerometer for 7 days (counts)
Adherence to the Mediterranean diet | 1 year
  Diet will be assessed with the Mediterranean Diet (MD) adherence questionnaire, developed in the PREDIMED project and consisting of 14 items with dichotomous responses.(points)
Sleep quality and quantity | 1 year
  Pittsburgh Sleep Quality Index (PSQI) which assesses the quality of sleep disturbance in the last month. It is composed of 19 items. The cut-off point for poor sleep quality is 5 points or higher. (points)
Sleep disruption | 1 year
  The Ford Insomnia Response to Stress Test, which assesses the likelihood of sleep disruption (points)

CONTACTS AND LOCATIONS:
Overall Officials: Manuel A Gomez-Marcos, Dr, Principal Investigator — Primary Care Research Unit
Locations (1):
- Primary Care Research Unit of Salamanca, Salamanca, Spain

IPD SHARING:
Plan to Share IPD: No